CLINICAL TRIAL: NCT03734627
Title: Gastrointestinal Nutrient Transit and Enteroendocrine Function After Upper Gastrointestinal Surgery
Acronym: EndoGut
Status: Completed | Type: Observational
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dr Jessie A Elliott, Clinical Research Fellow, St. James's Hospital, Ireland
Other Study IDs: CRFSJ075 and 0095; 2016-02-CA(9) (Other: SJH/AMNCH Research Ethics Committee); 2016-03-11(1) (Other: SJH/AMNCH Research Ethics Committee)
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Esophageal Cancer; Nutrition Disorders; Appetite Disorders; Dumping Syndrome; Delayed Gastric Emptying; Surgery
Keywords: Gut hormones; GLP-1; Enteroendocrine L-cell; Early satiety; Dumping syndrome; Gastrointestinal transit; Insulin; Octreotide; Somatostatin; Esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms; Nutrition Disorders; Feeding and Eating Disorders; Dumping Syndrome; Gastroparesis; Insulin Resistance | interventions — Octreotide; Saline Solution; Acetaminophen; Sulfasalazine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Plasma
  * Serum
  * Duodenal biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Upper Gastrointestinal Surgery - Transit
  Interventions: Drug: Octreotide Acetate; Drug: Saline Solution; Drug: Paracetamol; Drug: Sulfasalazine
- Control - Transit
  Interventions: Drug: Octreotide Acetate; Drug: Saline Solution; Drug: Paracetamol; Drug: Sulfasalazine
- Upper Gastrointestinal Surgery - Gut Function
  Interventions: Diagnostic Test: Duodenal biopsy
- Control - Gut Function
  Interventions: Diagnostic Test: Duodenal biopsy

INTERVENTIONS:
Drug: Octreotide Acetate — 50mcg octreotide acetate by subcutaneous injection 10 minutes prior to a 400kcal mixed meal challenge
  Groups: Control - Transit; Upper Gastrointestinal Surgery - Transit
Drug: Saline Solution — Equivalent volume of 0.9% saline by subcutaneous injection 10 minutes prior to a 400kcal mixed meal challenge
  Groups: Control - Transit; Upper Gastrointestinal Surgery - Transit
Drug: Paracetamol — Paracetamol 1g by mouth consumed with a 400kcal mixed meal challenge
  Groups: Control - Transit; Upper Gastrointestinal Surgery - Transit
Drug: Sulfasalazine — 1g sulfasalazine by mouth consumed with a 400kcal mixed meal challenge
  Groups: Control - Transit; Upper Gastrointestinal Surgery - Transit
Diagnostic Test: Duodenal biopsy — Biopsy from the second part of the duodenum taken at routine endoscopic surveillance, undertaken for another clinical indication.
  Groups: Control - Gut Function; Upper Gastrointestinal Surgery - Gut Function

SUMMARY:
The incidence of oesophagogastric cancer has increased by 400% since the 1970s in Ireland and the United Kingdom. In addition, refinement of perioperative management and the now widespread use of multimodal protocols for patients with locally advanced disease have significantly improved outcomes for patients with oesophagogastric cancer treatable with curative intent. Despite significant advances in chemoradiotherapy, surgical resection remains the primary curative option.

Unintentional weight loss and nutritional complications represent serious concerns for patients after radical resection, even among those who remain free from recurrent disease in the long-term. A study from the Swedish Esophageal and Cardia Cancer Registry reported a mean three year weight loss of 10.8% among disease-free patients, with 33.8% of this cohort demonstrating malnutrition at three years post-oesophagectomy.

Mechanisms contributing to weight loss for disease-free patients after upper gastrointestinal surgery are poorly understood, however an association between increasing magnitude of weight loss and the presence of increased satiety is described. Our recent studies at SJH have demonstrated four fold elevated postprandial satiety gut hormone concentrations after oesophagectomy, compared with baseline preoperative values. Postprandial gut hormone levels correlate significantly with postprandial symptoms and altered appetite at 3 months postoperatively, and with body weight loss at 2 years postoperatively. However, the mechanism leading to exaggerated postprandial gut hormone production after upper gastrointestinal surgery is poorly understood, limiting targeted therapeutic options.

In this study, we aim to characterise the role of altered nutrient transit and enteroendocrine cell function in the pathophysiology of excessive post-prandial gut hormone responses after upper gastrointestinal surgery. To do this, we will measure the gut hormone response to a standardised 400 kcal meal, as per previous studies, while concurrently assessing gastrointestinal transit time, and enteroendocrine cell morphology and function. In this way, we will determine whether the magnitude of the postprandial gut hormone response correlates with the rate of nutrient transit into the enteroendocrine L-cell rich small intestine, and whether enteroendocrine cell adaptation occurs after oesophagectomy.

Furthermore, we have previously observed that gut hormone suppression using octreotide is associated with increased ad libitum among subjects after upper gastrointestinal cancer surgery (Elliott JA et al, Annals of Surgery, 2015). The mechanism of action of octreotide may relate to SSTR-5-mediated negative feedback to the enteroendocrine L-cell, but this medication may additionally reduce enteroendocrine L-cell responses through its inhibitory effect on gastrointestinal motility - reducing the rapidity with which nutrients are delivered to the small intestine - and small intestinal nutrient sensing via inhibition of the Na+-dependent glucose transporter SGLT-18-10. Through conduction of this double-blind, randomised, placebo-controlled crossover study, we aim to establish the mechanism of action of octreotide-mediated increased food intake in patients after gastrointestinal surgery. This may inform the design of future targeted interventions for this patient group.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

1. History of upper gastrointestinal surgery at least 9 months previously

Control group:

1. Patients with suspected or confirmed non-dysplastic Barrett's oesophagus or reflux who are age, weight and gender matched to the patient cohort

Exclusion Criteria:

1. Pregnancy, breastfeeding
2. Recurrent disease after surgery
3. Other active malignancy
4. Significant psychiatric disorder or cognitive decline or communication impairment limiting capacity to provide informed consent
5. Other disease or medication which may impact gut hormone physiology
6. Previous upper gastrointestinal resection
7. Certain allergies or dietary intolerances
8. Anticoagulants

Patients with contraindications to the study medications (as per www.medicines.ie) will not be automatically excluded, but will be invited to participate in an attenuated protocol where that agent is not given. It is not anticipated that this will be a frequent occurrence, however this strategy will minimise unnecessary participant exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at least 9 months post upper gastrointestinal surgery and age-, weight- and sex-matched control subjects with gastroesophageal reflux disease or non-dysplastic Barrett's oeosophagus.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve for paracetamol at 30 minutes after a 400kcal mixed meal stimulus | 30 minutes post meal

SECONDARY OUTCOMES:
Peak paracetamol level | Within 300 minutes post meal
GLP-1 area under the curve over 300 minutes after a 400kcal mixed meal stimulus | Within 300 minutes post meal
Glucose area under the curve over 300 minutes after a 400kcal mixed meal stimulus | Within 300 minutes post meal
Insulin area under the curve over 300 minutes after a 400kcal mixed meal stimulus | Within 300 minutes post meal
Visual analogue scales | Within 300 minutes post meal
EORTC health related quality of life | At one year post surgery, on the day of assessment

OTHER OUTCOMES:
Duodenal enteroendocrine cell density | At one year post surgery, on the day of assessment
Duodenal enteroendocrine L-cell density | At one year post surgery, on the day of assessment
Duodenal enteroendocrine cell mRNA expression profile | At one year post surgery, on the day of assessment

CONTACTS AND LOCATIONS:
Overall Officials: John V Reynolds, MD FRCS, Principal Investigator — St. James's Hospital, Dublin, Ireland; Carel W le Roux, FRCP FRCPath PhD, Principal Investigator — Conway Institute of Biomolecular and Biomedical Research
Locations (2):
- Ireland (2):
  - Department of Surgery, St. James's Hospital, Dublin
  - Wellcome Trust-Health Research Board Clinical Research Facility, St. James's Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott JA, Docherty NG, Eckhardt HG, Doyle SL, Guinan EM, Ravi N, Reynolds JV, Roux CWL. Weight Loss, Satiety, and the Postprandial Gut Hormone Response After Esophagectomy: A Prospective Study. Ann Surg. 2017 Jul;266(1):82-90. doi: 10.1097/SLA.0000000000001918. PMID 27455150
- [Background] Elliott JA, Jackson S, King S, McHugh R, Docherty NG, Reynolds JV, le Roux CW. Gut Hormone Suppression Increases Food Intake After Esophagectomy With Gastric Conduit Reconstruction. Ann Surg. 2015 Nov;262(5):824-29; discussion 829-30. doi: 10.1097/SLA.0000000000001465. PMID 26583672